CLINICAL TRIAL: NCT04552899
Title: A Phase III Randomized, Double-blind, Placebo Controlled Trial to Evaluate the Efficacy and Safety of PRM-151 in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: A Study to Evaluate the Efficacy and Safety of Recombinant Human Pentraxin-2 (rhPTX-2; PRM-151) in Participants With Idiopathic Pulmonary Fibrosis
Acronym: STARSCAPE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated by Sponsor as the futility analysis outcome indicated that the study was unlikely to meet the predefined primary objective of the study. No new safety concerns were identified.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WA42293; 2020-000791-38 (EudraCT Number)
Record Dates: First submitted 2020-09-14; First posted 2020-09-17 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-03

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — PRM-151

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Zinpentraxin Alfa (Experimental): Participants will receive intravenous (IV) infusions of Zinpentraxin Alfa over 50-70 minutes on Days 1, 3 and 5, then followed by infusions every 4 weeks (Q4W) to Week 48.
  Interventions: Drug: PRM-151 (Zinpentraxin Alfa)
- Placebo (Placebo Comparator): Participants will receive IV infusions of placebo over 50-70 minutes on Days 1, 3 and 5, followed by infusions Q4W to Week 48.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PRM-151 (Zinpentraxin Alfa) — A 10 mg/kg IV infusion of PRM-151 based on the participants weight will be administered on Days 1, 3 and 5 followed by infusions Q4W to Week 48.
  Arms: Zinpentraxin Alfa
Drug: Placebo — Placebo matching PRM-151 will be administered by IV infusion on Days 1, 3 and 5, followed by infusions Q4W to Week 48.
  Arms: Placebo

SUMMARY:
This phase III study will evaluate the efficacy, safety and pharmacokinetics (PK) of recombinant human pentraxin-2 (rhPTX-2; PRM-151) zinpentraxin alfa, compared with placebo in participants with idiopathic pulmonary fibrosis (IPF).

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of IPF per the 2018 American Thoracic Society (ATS)/European Respiratory Society (ERS)/Japanese Respiratory Society (JRS)/Latin American Thoracic Society (ALAT) Clinical Practice Guideline
* High-resolution computed tomography (HRCT) pattern consistent with the diagnosis of IPF, confirmed by central review of Chest HRCT and central review of any available lung biopsy (LB)
* Minimum 6 minute walk distance (6MWD) of 150 meters with maximum use of 6 L/min at sea-level and up-to 8 L/min at altitude of supplemental oxygen while maintaining oxygen saturation of greater than or equal to (>/= )83% during the 6 minute walk test (6MWT) during screening
* FVC >/= 45% predicted during screening as determined by the over-reader
* Forced expiratory volume in 1 second (FEV1)/FVC ratio greater than (>) 0.70 during screening determined by the over-reader
* Diffusing capacity for carbon monoxide (DLCO) >/= 30% and less than or equal to (</=) 90% of predicted at screening as determined by the over-reader
* If receiving pirfenidone or nintedanib treatment for IPF, the participant must have been on treatment for at least 3 months and a stable dose for at least 4 weeks prior to screening, and during screening
* If not currently receiving nintedanib or pirfenidone treatment (either treatment naïve or having previously taken and discontinued) must have discontinued such treatment >/= 4 weeks prior to screening and during screening
* Anticipated life expectancy of at least 12 months at baseline
* Participant and investigator considered all medicinal treatment options and/or possibly lung transplantation prior to considering participation in the study.
* For women of childbearing potential (excluding participant enrolling in Japan): agreement to remain abstinent or use contraception
* For men: agreement to remain abstinent or use a condom, and agreement to refrain from donating sperm
* Anticipated life expectancy of at least 12 months at baseline, according to the investigator's judgment
* For participant enrolled in the extended China enrollment phase: current resident of mainland China, Hong Kong, or Taiwan, and of Chinese ancestry

Exclusion Criteria:

* Evidence of other known causes of Interstitial Lung Disease (ILD)
* FVC% predicted value showing repeated increase in the 6 months period prior to screening and including screening value
* Emphysema present on greater than or equal to (>/=) 50% of the HRCT, or the extent of emphysema is greater than the extent of fibrosis, according to central review of the HRCT
* Receiving nintedanib in combination with pirfenidone
* Received cytotoxic, immunosuppressive, cytokine modulating, or receptor antagonist agents (including but not limited to methotrexate, azathioprine, mycophenolate mofetil, cyclophosphamide, cyclosporine or other steroid sparing agent) within 4 weeks prior to or during screening
* Receiving systemic corticosteroids equivalent to prednisone > 10 mg/day or equivalent within 2 weeks prior to or during screening
* Acute respiratory or systemic bacterial, viral, or fungal infection either during screening or prior to screening and not successfully resolved 4 weeks prior to screening visit
* Participants with active or latent tuberculosis (confirmed within the 6 months prior to or during screening, by a positive screening test [interferon gamma release assay])
* Resting oxygen saturation of < 89% using up to 4 L/min of supplemental oxygen at sea level and up to 6 L/min at altitude (>/= 5000 feet [1524 meters] above sea level) during screening
* Class IV New York Heart Association chronic heart failure
* Historical evidence of left ventricular ejection fraction < 35%
* Presence of pulmonary hypertension that, in the investigator's opinion, would substantially limit the ability to comply with study requirements or may influence any of the safety or efficacy assessments included in the study
* Cardiopulmonary rehabilitation program based on exercise training that has been completed within 8 weeks prior to screening or planned to start during the participant enrollment in this trial
* History of smoking, alcohol or substance abuse disorder, or a malignancy
* Previous treatment with PRM-151
* Clinically significant abnormality on ECG during screening that, in the opinion of the investigator, may pose an additional risk in administering study drug to the participant including prolonged corrected QT interval > 450 ms (for men) or > 470 ms (for women) on ECG during screening based on the Fridericia correction formula
* Clinically significant laboratory test abnormalities during screening (hematology, serum chemistry, and urinalysis) that, in the opinion of the investigator, may pose an additional risk in administering study drug to the participant
* Pregnant or breastfeeding, or become pregnant during the study or within 8 weeks after the final dose of PRM-151
* Women of childbearing potential (Only for participants enrolling in Japan)

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 665 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (360):
- United States (72):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner University Medical Center Phoenix; Main Pharmacy, Phoenix, Arizona
  - Lovelace Scientific Resources, Inc., Phoenix, Arizona
  - UC Irvine Medical Center, Orange, California
  - Stanford Hospital and Clinics, Palo Alto, California
  - University of California Davis, Sacramento, California
  - Inst. of Healthcare Assessment, Inc., San Diego, California
  - UCSF Medical Center, San Francisco, California
  - Paloma Medical Group, San Juan Capistrano, California
  - William Sansum Diabetes Center, Santa Barbara, California
  - University of Colorado - Anschutz Medical Campus (University of Colorado Health Sciences Center), Aurora, Colorado
  - National Jewish Health Medical Center, Denver, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Meris Clinical Research, Brandon, Florida
  - Florida Lung, Asthma and Sleep Specialists (FLASS) - Celebration, Celebration, Florida
  - Advanced Pulmonary & Sleep Research Institute of Florida, Daytona Beach, Florida
  - University of Florida Division of Pulmonary, Critical Care, and Sleep Medicine, Gainesville, Florida
  - Malcom Randall VA Medical Center, Gainesville, Florida
  - University of Florida Health Pulmonology - Jacksonville, Jacksonville, Florida
  - Advanced Pulmonary Research Institute, Loxahatchee Groves, Florida
  - San Marcus Research Clinic Inc., Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Central Florida Pulmonary Group, PA, Orlando, Florida
  - Sarasota Memorial Health Care System; Cancer Research Program, Sarasota, Florida
  - University of South Florida, Tampa, Florida
  - Integral ? Clinical Trial Solutions, Weston, Florida
  - Clinical Site Partners Orlando, Winter Park, Florida
  - Emory University, Atlanta, Georgia
  - Piedmont Healthcare Pulmonary and Critical Care Research, Austell, Georgia
  - NorthShore University HealthSystem, Evanston, Illinois
  - Indiana Univ School of Med, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics; Investigational Drug Services, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville Health Sciences Center, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women'S Hospital, Boston, Massachusetts
  - Covenant Medical Center - Cooper, Saginaw, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - The Lung Research Center, Chesterfield, Missouri
  - Washington University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Pulmonary & Allergy Associates, Summit, New Jersey
  - Lenox Hill Hospital, New York, New York
  - American Health Research Inc., Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Pulmonix Research, Greensboro, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Mercy St. Vincent Medical Center, Toledo, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Jefferson University Physicians (JUP) - Jefferson Pulmonary, Philadelphia, Pennsylvania
  - Temple University Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina Hospital, Charleston, South Carolina
  - SleepMed of South Carolina, Columbia, South Carolina
  - Lowcountry Lung and Critical Care, North Charleston, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Horizon Clinical Research Group, Cypress, Texas
  - Cardiopulmonary Research Science and Technology Institute, Dallas, Texas
  - University of Texas Southwestern Medical Center; Heart and Lung Clinic, Dallas, Texas
  - University of Texas Medical Branch; Cardiology Department, Galveston, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Metroplex Pulmonology & Sleep Center, McKinney, Texas
  - Audie L. Murphy VA Hospital, STVHCS, San Antonio, Texas
  - University Of Utah Hosp & Clin; Investigational Pharmacy, Salt Lake City, Utah
  - Inova Fairfax Hospital/IHVI; Cardiology, Falls Church, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Wisconsin-Madison, Madison, Wisconsin
- Argentina (8):
  - Hospital Britanico de Buenos Aires, Ciudad Autonoma Buenos Aires
  - Fundacion Respirar (Centro Medico Dra. De Salvo), Ciudad Autonoma Buenos Aires
  - Instituto de Medicina Respiratoria, IMeR; Clinic/Outpatient Facility, Córdoba
  - Centro Medico de Enfermedades Respiratorias (CEMER), Florida, Buenos Aires
  - Centro de estudios respiratorios, Mar del Plata
  - Fundacion Scherbovsky, Mendoza
  - INSARES, Mendoza, Mendoza City
  - Investigaciones en Patologias Respiratorias, San Miguel de Tucumán
- Australia (9):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Cairns Base Hospital; Cancer Care Centre, Cairns, Queensland
  - Lung Research Queensland, Nundah, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - The Queen Elizabeth Hospital, Adelaide, South Australia
  - Austin Hospital; Cancer Clinical Trials Centre, Melbourne, Victoria
  - Monash Medical Centre; Medicine, Melbourne, Victoria
  - The Alfred Hospital, Prahan, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Austria (2):
  - Klinikum Klagenfurt am Wörthersee; 2. Medizinische Abteilung, Klagenfurt
  - Landeskrankenhaus Salzburg; Gynäkologie Und Onkologie, Salzburg
- Belgium (5):
  - ULB Hôpital Erasme, Brussels
  - Cliniques Universitaires Saint-Luc; Pharmacy, Brussels
  - UZ Leuven, Leuven
  - C. H. U. Sart-Tilman; Laboratory, Liège
  - CHU UCL Namur / site Godinne, Yvoir
- Brazil (2):
  - Hospital das Clinicas - UFMG, Belo Horizonte, Minas Gerais
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
- Canada (10):
  - University of Alberta Hospital, Edmonton, Alberta
  - Synergy Respiratory Care, Sherwood Park, Alberta
  - Kelowna Respiratory and Allergy Clinic, Kelowna, British Columbia
  - Vancouver General Hospital; Gordon and Leslie Diamond Health Care, Vancouver, British Columbia
  - Eastern Health - General Hospital, St. John's, Newfoundland and Labrador
  - The Rhema Research Institute, Owen Sound, Ontario
  - Dr. Syed Anees Medicine Profession Corporation, Windsor, Ontario
  - Centre Hospitalier de l'Universite de Montreal - Notre - Dame Hos pital, Montreal, Quebec
  - McGill University, Montreal Chest Institute; Viral and other Infectious, Montreal, Quebec
  - C.I.C. Mauricie, Trois-Rivières, Quebec
- China (31):
  - CMU-Beijing Chao-Yang Hospital-Beijing Institute of Respiratory Medicine, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Beijing Friendship Hospital Affiliated of Capital University of Medical Science, Beijing
  - Peking University Third Hospital, Beijing
  - Peking Union Medical College Hospital; Pharmacy, Beijing
  - Xiangya Hospital Central South University, Changsha
  - The Second Xiangya Hospital of Central South University, Changsha
  - The Third Xiangya Hospital Of Central South University, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - Southern Medical University Nanfang Hospital, Guangdong Province Guangzhou City
  - The First Affilicated Hospital, Sun Yat-sen University, Guangzhou
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - 1st Affiliated Hospital of Zhejiang University; Clinical Trial Pharmacy, Hangzhou
  - Inner Mongolia Autonomous Region People's Hospital, Hohhot
  - Qilu Hospital of Shandong University, Jinan
  - The 1st Affiliated Hospital of Nanchang Unversity, Nanchang
  - Nanjing Drum Tower Hospital, the Affiliated Hospital of Nanjing University Medical School, Nanjing
  - Ningbo First Hospital, Ningbo
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai
  - Huadong Hospital Affiliated to Fudan University, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - China Medical University (CMU) First Affiliated Hospital, Shenyang
  - Shengjing Hospital of China Medical University, Shenyang
  - Hebei Medical University - The Second Hospital, Shijiazhuang
  - Tianjin Medical University General Hospital, Tianjin
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Wuxi People's Hospital, Wuxi
  - Tangdu Hospital, The Fourth Military Medical University; Neurology Department, Xi'an
  - Qinghai Provincial People?s Hospital, Xining
  - Henan University of Traditional Chinese Medicine (HUTCM) The First Affiliated Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
- Czechia (6):
  - Fakultní Nemocnice Brno, Brno
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni Nemocnice Plzen - Klinika Pneumologie a Ftizeologie, Pilsen
  - Thomayerova nemocnice; Lekarna - pavilon H, Prague
  - Nemocnice Na Bulovce, Prague
  - Krajská nemocnice T. Bati, a. s., Zlín
- Denmark (3):
  - Aarhus Universitetshospital Skejby, Aarthus N
  - Gentofte Hospital, Hellerup
  - Odense Universitetshospital, Odense C
- Turku University Hospital, Turku, Finland
- France (16):
  - Hopital Avicenne, Bobigny
  - Centre Hospitalier Regional Universitaire de Brest - Hopital de la Cavale Blanche, Brest
  - Hopital Louis Pradel, Bron
  - Hospital d Instructions des Armees Percy, Clamart
  - CHU Dijon Bourgogne Hôpital François Mitterand, Dijon
  - CHU de Grenoble - Hôpital André Michallon; Pole Pharmacie, La Tronche
  - Centre Hospitalier Regional Universitaire de Lille, Lille
  - Servie de Pneumologie et centre de Transplantation Pulmonaire, Marseille
  - CHU de Montpellier Hopital Arnaud de Villeneuve; de Génétique, Montpellier
  - CHU Nice - Hôpital Pasteur 2, Nice
  - Hopital Bichat Claude Bernard; CIC, Paris
  - European Hospital Georges Pompidou (HEGP), Paris
  - Hopital Haut Leveque, Pessac
  - Centre Hospitalier Universitaire de Reims; l'Hopital Maison Blanche, Reims
  - CHU de Rennes - Hopital de Pontchaillo, Rennes
  - CHU Tours - Hôpital Bretonneau; Pharmacie, Tours
- Germany (14):
  - Zentralklinik Bad Berka GmbH; Pneumologie, Bad Berka
  - Evang. Lungenklinik Berlin Klinik für Pneumologie, Berlin
  - Universitatsklinikum Essen; Innere Klinik, Essen
  - IFS - Interdisziplinäres Facharztzentrum; Institut für klinische Forschung Pneumologie, Frankfurt am Main
  - Universitatsklinikum Gießen und Marburg GmbH, Giessen
  - Medizinische Hochschule Hannover; Zentrum Innere Medizin - Klinik fur Pneumologie, Hanover
  - Thoraxklinik-Heidelberg gGmbH; Apotheke der Thoraxklinik, Heidelberg
  - Universitätsklinikum des Saarlandes; Klinik für Augenheilkunde, Homburg/Saar
  - Lungenfachklinik Immenhausen, Immenhausen
  - Universitatsklinikum Leipzig; Apotheke, Leipzig
  - IKF Pneumologie Mainz Helix Medical Excellence Center Mainz, Mainz
  - Praxis für Pneumologie Dr. Silke Mronga & Dr. Lukas Jerrentrup, Marburg
  - Lungenklinik Münnerstadt, Thoraxzentrum Bezirk Unterfranken, Münnerstadt
  - Krankenhaus Bethanien gGmbH, Solingen
- Greece (9):
  - Evangelismos Hospital; Department of Critical Care and Pulmonary Services, Athens
  - Attikon University General Hospital, Chaïdári
  - University General Hospital of Heraklion, Heraklio
  - University Hospital of Ioannina; Pulmonology Department, Ioannina
  - Hospital is University General Hospital of Larissa, Larissa
  - Athens Medical Center, Marousi
  - University General Hospital of Patras, Pátrai
  - "General hospital of Chest Diseases ""Sotiria"", 7th Pulmonary Clinic ", Sotiria Athens
  - General Hospital of Thessaloniki G. Papanikolaou, Thessaloniki
- Hong Kong (2):
  - Prince of Wales Hospital; Dept. of Medicine & Therapeutics, Hong Kong
  - The University of Hong Kong; Queen Mary Hospital, Hong Kong
- Hungary (5):
  - Semmelweis University, Budapest
  - Debreceni Egyetem, Debrecen
  - Markusovszky Egyetemi Oktatokorhaz ; SZEMESZET, Szombathely
  - Szent Borbala Korhaz, Tatabánya
  - Tudogyogyintezet Torokbalint; Onkologiai és Jarobeteg Centrum, Törökbálint
- Israel (14):
  - Barzilai Medical Center; Neurology Department, Ashkelon
  - Ben-Gurion University of the Negev - Soroka University Medical Center - Pulmonology Institute, Beersheba
  - Shamir medical center, Be’er Ya‘aqov
  - Rambam Health Care Campus, Haifa
  - Bnai Zion Medical Center; Internal Medicine, Haifa
  - Carmel Medical Center; Obstetrics and Gynecology, Haifa
  - Edith Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center; Nrphrology Dept., Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petach Tiqwa
  - The Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Tel-Aviv Sourasky Medical Center; Department of Pulmonary, Tel Aviv
- Italy (28):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo, Abruzzo
  - Policlinico Riuniti di Foggia - Department of Medical and Surgical Sciences - University of Foggia, Foggia, Apulia
  - Ospedale di Ostuni - Pneumologia, Ostuni, Apulia
  - AORN Ospedali dei Colli Ospedale Monaldi; UOC Pneumologia ad indirizzo Oncologico, Napoli, Campania
  - Azienda Ospedaliera Dei Colli, Napoli, Campania
  - Azienda Ospedaliera Universitaria Federico II, Napoli, Campania
  - Università degli Studi di Napoli Federico II; Dipartimento di Scienze Oftalmologiche, Napoli, Campania
  - Ospedale Morgagni Pierantoni; Patologia clinica, Forlì, Emilia-Romagna
  - A.O.U. Policlinico di Modena, Modena, Emilia-Romagna
  - Azienda Sanitaria Universitaria Integrata di Trieste, Trieste, Friuli Venezia Giulia
  - Policlinico Tor Vergata - U.O.C. Malattie Apparato Respiratorio, Rome, Lazio
  - Fondazione Policlinico Universitario A Gemelli; Servizio di Farmacia, Rome, Lazio
  - "Asst Rhodense - Unità operativa di pneumologia Ospedale ""Guido Salvini"" ", Garbagnate Milanese, Lombardy
  - Ospedale San Giuseppe; U.O. di Pneumologia, Milan, Lombardy
  - Asst Santi Paolo E Carlo, Milan, Lombardy
  - Ospedale San Gerardo, Monza, Lombardy
  - Fondazione IRCCS Policlinico San Matteo Divisione di EmatologiaDipartimento di Onco-Ematologia, Pavia, Lombardy
  - A.O.U. S. Luigi Gonzaga; Interstiziopatie Malattie Rare Polmone, Orbassano (TO), Piedmont
  - Azienda Ospedaliera Universitaria Citta della Salute e della Scienza di Torino; Ospedale Molinette, Turin, Piedmont
  - A.O.U. Sassari; Dip. Medicina Clinica e Sperimentale, Sassari, Sardinia
  - Azienda Ospedaliero - Universitaria Policlinico - Vittorio Emanuele, Catania, Sicily
  - Az. Osp. Univ. P. Giaccone; UOC di Pneumologia, Palermo, Sicily
  - Ismett Istituto Mediterraneo Trapianti E Terapie Alta Specializzazione;Pneumologia, Palermo, Sicily
  - Azienda Ospedaliero Universitaria Ospedali Riuniti, Torrette Di Ancona, The Marches
  - AOUC Azienda Ospedaliero-Universitaria Careggi; Neurologia 2, Florence, Tuscany
  - A.O. Univ. Senese Policlinico S. Maria alle Scotte; Dip. Medicina clinica e Scienze Immunologiche, Siena, Tuscany
  - Azienda Ospedale Università Di Padova; Clinica Pneumologica, Padua, Veneto
  - University of Padova Ca' Foncello Hospital Immunologic & Respiratory Rare Diseases Center, Treviso, Veneto
- Japan (20):
  - Nagoya University Hospital, Aichi
  - Chiba University Hospital, Chiba
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Fukuoka University Hospital, Fukuoka
  - Kobe City Medical Center General Hospital, Hyōgo
  - National Hospital Organization Himeji Medical Center, Hyōgo
  - Kameda Medical Center, Kamogawa
  - Kanagawa Cardiovascular and Respiratory Center, Kanagawa
  - Nippon Medical School Musashi Kosugi Hospital, Kawasaki-Shi
  - Saiseikai Kumamoto Hospital, Kumamoto
  - Nagasaki University Hospital, Nagasaki
  - National Hospital Organization Ibarakihigashi National Hospital; Center for Clinical Research, Naka-gun
  - Kurashiki Central Hospital, Okayama
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Sakaishi
  - Tosei General Hospital, Seto-shi
  - Tenri Hospital, Tenri-Shi
  - Jichi Medical University Hospital, Tochigi
  - Tokushima University Hospital, Tokushima
  - Tokyo Medical Ando Dentaluni Hospital Faculty of Medicine; Surgical Oncology, Tokyo
  - Center Hospital of the National Center for Global Health and Medicine, Tokyo
- Mexico (5):
  - INER- Instituto Nacional de Enfermedades Respiratorias"Ismae, Mexico City, Mexico CITY (federal District)
  - Centro Respiratorio de México, México, Mexico CITY (federal District)
  - Unidad Médica para la Salud Integral UMSI, San Nicolás de los Garza, Nuevo León
  - Unidad de Investigacion CIMA SC, Chihuahua City
  - CICC Morelia, Morelia
- Netherlands (3):
  - VU Medisch Centrum, Amsterdam
  - Sint Antonius Ziekenhuis, locatie Nieuwegein, Nieuwegein
  - Erasmus Medisch Centrum, Rotterdam
- New Zealand (5):
  - Auckland City Hospital, Auckland
  - NZ Respiratory & Sleep Institute, Auckland
  - University of Otago, Christchurch, Christchurch
  - Waikato Hospital; Gastro Research, Hamilton
  - Tauranga Hospital, Tauranga
- Norway (3):
  - Helse Bergen HF Haukeland universitetssykehus, Bergen
  - Akershus universitetssykehus, Lørenskog
  - Oslo University Hospital HF, Rikshospitalet, Oslo
- Poland (3):
  - Centrum Medycyny Oddechowej Mroz sp. j., Bia?ystok
  - Nasz Lekarz Osrodek Badan Klinicznych, Bydgoszcz
  - Uniwersytecki Szpital Kliniczny Nr 1 im.N.Barlickiego Oddzial Kliniczny Pneumonologii i Alergologii, Lodz
- Portugal (8):
  - Hospital de Braga; Centro Clínico Académico (Piso 1, Ala E), Braga
  - Centro Hospitalar Algarve, Faro
  - Hospital Senhora da Oliveira ? Guimarães, E.P.E, Guimarães
  - Centro Hospitalar Universitario Lisboa Norte - Hospital Pulido Valente, Lisbon
  - Centro Hospitalar do Porto - Hospital de Santo António, Porto
  - Hospital de Sao Joao; Centro de Investigacao, Porto
  - Hospital de Santa Luzia, Porto
  - CHVNG/E_Unidade 1; Servico de Pneumologia, Vila Nova de Gaia
- Singapore (2):
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital; Oncology, Singapore
- South Africa (2):
  - University of Cape Town Lung Institute; Lung Clinical Research, Cape Town
  - Vergelegen Medi-Clinic, Somerset West
- South Korea (11):
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - The Catholic University of Korea Bucheon St. Mary's Hospital, Gyeonggi-do
  - Gacheon University Gil Medical Center, Namdong-gu
  - Seoul National University Bundang Hospital, Seongnam-si
  - The Catholic University of Korea Yeouido St. Mary's Hospital; Hematology-Oncology, Seoul
  - Seoul National University Hospital (SNUH) - Medical Oncology Center, Seoul
  - Soonchunhyang University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - The Catholic University of Korea Seoul St. Mary?s Hospital, Seoul
- Spain (30):
  - Hospital Txagorritxu, Vitoria-Gasteiz, Alava
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Parc Taulí Sabadell Hospital Universitari, Sabadell, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Complexo Hospitalario Universitario de Santiago (CHUS) - Hospital Clinico Universitario, Santiago de Compostela, LA Coruña
  - Hospital Universitario del Henares, Coslada, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Universidad de Navarra - Clinica Universitaria de Navarra (CUN), Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario de Canarias, S. Cristobal de La Laguna, Tenerife
  - Hospital Galdakao-Usansolo, Galdakao, Vizcaya
  - Hospital de la Santa Creu i Sant Pau; Servicio de Neumologia, Barcelona
  - Vall d?Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona
  - Hospital Virgen de las Nieves; Servicio de Neumologia, Granada
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario La Paz, Madrid
  - Clínica Universidad de Navarra ? Madrid, Madrid
  - Hospital Ramón y Cajal;Servicio de Neumología, Madrid
  - Hosp. Clinico San Carlos, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz., Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Arnau de Vilanova (Valencia), Valencia
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Skånes universitetssjukhus Malmö, Malmo, Sweden
- Switzerland (2):
  - Inselspital Bern Universitätsklinik für Pneumologie, Bern
  - Hopital Neuchatelois Pourtales (Hopitaux Cadolles Pourtales), Neuchâtel
- Taiwan (7):
  - Buddhist Tzu Chi Dalin General Hospital; Rheumatology, Chiayi City
  - Kaohsiung Medical University Hospital; Chung-Ho Memorial Hospital, Kaoshiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Far Eastern Memorial Hospital; Department of Clinical Pathology, Taipei
  - Veterans General Hospital - Taichung, Xitun Dist.
- Turkey (Türkiye) (14):
  - Istanbul Universitesi Onkoloji Enstitüsü Hastanesi, ?stanbul
  - Cukurova Universitesi Tip Fakultesi Balcali Hastanesi; Balcali, Adana
  - Ankara Universitesi Tip Fakultesi Hastaneleri - Cebeci Hastanesi, Ankara
  - Uludag Universitesi - Saglik Uygulama ve Arastirrma Merkezi, Bursa
  - Gaziantep Universitesi - Sahinbey Arastirma ve Uygulama Hastanesi, Gaziantep
  - Yedikule Gogus Hastaliklari ve Gogus Cerrahisi EAH;Gogus Hastaliklari, Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi, Izmir
  - Dokuz Eylul University Faculty of Medicine; Chest Diseases, Izmir
  - Erciyes Üniversitesi T?p Fakültesi, Kayseri
  - Kocaeli Universitesi Tip Fakultesi, Kocaeli
  - Marmara Universitesi Hastanesi Marmara University Hospital, Maltepe
  - Mersin Üniversitesi Tip Fakültesi, Mersin
  - Akdeniz University Faculty of Medicine Department of Pulmonology, Muratpasa/Antalya
  - Koc Universitesi (KU) Tip Fakultesi (Koc University School of Medicine), Sarıyer
- Ukraine (3):
  - Municipal Non-Profit Enterprise City Clinical Hospital #16 of Dnipro City Council, Dnipro, Katerynoslav Governorate
  - National Academy of Medical Science of Ukraine (NAMS); NRCRM, Kyiv, KIEV Governorate
  - Yanovskyy Inst of Phth. & Pulm; Clinical-functional, Kyiv
- United Kingdom (4):
  - Edinburgh Royal Infirmary; Respiratory Department, Edinburgh
  - Royal Brompton Hospital; Respiratory Department, London
  - Manchester University NHS Foundation Trust - Wythenshawe Hospital, Manchester
  - North Manchester General Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/).
  For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Cong M, Carvalho Gontijo Weber R, Sakane S, Zhang V, Jiang C, Taura K, Kodama Y, DeMinicis S, Ganguly S, Brafman D, Chien S, Kramer M, Lupher M, Brenner DA, Xu J, Kisseleva T. Serum amyloid P (PTX2) attenuates hepatic fibrosis in mice by inhibiting the activation of fibrocytes and HSCs. Hepatol Commun. 2024 Oct 17;8(11):e0557. doi: 10.1097/HC9.0000000000000557. eCollection 2024 Nov 1. PMID 39761005
- [Derived] Richeldi L, Schiffman C, Behr J, Inoue Y, Corte TJ, Cottin V, Jenkins RG, Nathan SD, Raghu G, Walsh SLF, Jayia PK, Kamath N, Martinez FJ. Zinpentraxin Alfa for Idiopathic Pulmonary Fibrosis: The Randomized Phase III STARSCAPE Trial. Am J Respir Crit Care Med. 2024 May 1;209(9):1132-1140. doi: 10.1164/rccm.202401-0116OC. PMID 38354066
- [Derived] Mantovani A, Garlanda C. Humoral Innate Immunity and Acute-Phase Proteins. N Engl J Med. 2023 Feb 2;388(5):439-452. doi: 10.1056/NEJMra2206346. No abstract available. PMID 36724330

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 665 participants were enrolled across 275 investigative sites in 29 countries.
Pre-assignment Details: One participant who failed screening was enrolled in error and did not subsequently enter the study.
Groups:
- Zinpentraxin Alfa: Participants received intravenous (IV) infusions of Zinpentraxin Alfa over 50-70 minutes on Days 1, 3 and 5, then followed by infusions every 4 weeks (Q4W) to Week 48.
- Placebo: Participants received IV infusions of placebo over 50-70 minutes on Days 1, 3 and 5, followed by infusions Q4W to Week 48.
Period: Overall Study
Arm/Group | Zinpentraxin Alfa | Placebo
Started | 331 | 333
No Treatment (Participants who were randomized but didn't receive any treatment.) | 1 | 3
Completed | 56 | 49
Not Completed | 275 | 284
Not completed — Adverse Event | 4 | 3
Not completed — Death | 4 | 4
Not completed — Lost to Follow-up | 8 | 13
Not completed — Lung Transplant | 4 | 3
Not completed — Participant and physician wanted to withdraw participant from study | 0 | 1
Not completed — Physician Decision | 3 | 4
Not completed — Study Terminated By Sponsor | 237 | 239
Not completed — Withdrawal by Subject | 15 | 17

BASELINE CHARACTERISTICS:
Population: The randomized population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Zinpentraxin Alfa | Placebo | Total
Number analyzed (Participants) | 331 | 333 | 664
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.8 (7.3) | 70.6 (7.6) | 70.7 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 70 | 131
  Male | 270 | 263 | 533
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 27 | 47
  Not Hispanic or Latino | 302 | 299 | 601
  Unknown or Not Reported | 9 | 7 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 52 | 56 | 108
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 274 | 270 | 544
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Forced Vital Capacity (FVC [mL])
Time Frame: From Baseline up to Week 52
Population: The full analysis set included all randomized participants who received at least one administration (full or partial dose) of study drug and used the grouping according to the treatment assignment at randomization.
Measure: Mean (95% Confidence Interval); unit: Milliliters (mL)
Arm/Group | Zinpentraxin Alfa | Placebo
Number analyzed (Participants) | 330 | 330
Milliliters (mL) | -235.72 [-283.07 to -188.4] | -214.89 [-262.44 to -167.3]
Statistical Analysis 1: Comparison: Zinpentraxin Alfa vs Placebo; Test type: Superiority; p = 0.54, RCRM; Random Coefficient Regression Model (RCRM); Difference in Change from Baseline = -20.83, 95% CI 2-sided [-87.94 to 46.29], Standard Error of Mean 34.11

2. Secondary Outcome: Absolute Change in 6-minute Walk Distance (6MWD)
Time Frame: From Baseline up to Week 52
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Meters (m)
Arm/Group | Zinpentraxin Alfa | Placebo
Number analyzed (Participants) | 330 | 330
Meters (m) | -33.64 [-48.71 to -18.57] | -24.19 [-39.29 to -9.10]

3. Secondary Outcome: Absolute Change in FVC% Predicted
Time Frame: From Baseline up to Week 52
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Percent predicted
Arm/Group | Zinpentraxin Alfa | Placebo
Number analyzed (Participants) | 330 | 330
Percent predicted | -6.22 [-7.46 to -4.98] | -5.72 [-6.96 to -4.47]

4. Secondary Outcome: Time to Disease Progression
Time Frame: From Baseline up to 1 year
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Zinpentraxin Alfa | Placebo
Number analyzed (Participants) | 330 | 330
Months | 6.6 [5.6 to 9.1] | 8.2 [6.5 to 10.9]
Statistical Analysis 1: Comparison: Zinpentraxin Alfa; Test type: Superiority; p = 0.2512, Log Rank; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.91 to 1.47]

5. Secondary Outcome: Time to First Respiratory-related Hospitalizations
Time Frame: From Baseline up to 1 year
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Zinpentraxin Alfa | Placebo
Number analyzed (Participants) | 330 | 330
Months | NA [NA to NA] — NA = Not enough events available for estimation. | NA [NA to NA] — NA = Not enough events available for estimation.
Statistical Analysis 1: Comparison: Zinpentraxin Alfa; Test type: Superiority; p = 0.9833, Log Rank; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.51 to 1.97]

6. Secondary Outcome: Change in University of California, San Diego-Shortness of Breath Questionnaire (UCSD-SOBQ)
Description: The UCSD-SOBQ is a 24-item questionnaire used to assess dyspnea severity during specific activities (21 items) and limitations caused by dyspnea in daily life (4 items). Items are assessed using a 6-point scale. Total scores, once summed, can range from 0-120 with a higher score reflecting greater dyspnea severity.
Time Frame: At Baseline, Week 12, Week 24, Week 36 and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Zinpentraxin Alfa | Placebo
Number analyzed (Participants) | 276 | 271
Score on a scale
  Baseline | 28.9 (22.2) | 29.9 (22.6)
  Week 12: number analyzed (Participants) | 147 | 151
  Week 12 | 0.8 (13.0) | 4.0 (17.4)
  Week 24: number analyzed (Participants) | 106 | 110
  Week 24 | 3.2 (16.0) | 4.7 (16.8)
  Week 36: number analyzed (Participants) | 97 | 96
  Week 36 | 5.4 (17.5) | 6.9 (17.7)
  Week 52: number analyzed (Participants) | 37 | 35
  Week 52 | 11.1 (21.2) | 4.8 (14.8)

7. Secondary Outcome: Change in St. George Respiratory Questionnaire (SGRQ) Total Score
Description: The SGRQ is a 50-item respiratory-specific quality-of-life questionnaire. The questions assess the impact of disease on activity, functionality and symptoms. Each scale is scored from 0-100. A total score represents the weighted average of these three subscores. A lower score indicates best health while a higher score indicates worst health.
Time Frame: At Baseline, Week 12, Week 24, Week 36 and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Zinpentraxin Alfa | Placebo
Number analyzed (Participants) | 299 | 299
Score on a scale
  Baseline | 36.73 (18.63) | 37.66 (18.45)
  Week 12: number analyzed (Participants) | 172 | 179
  Week 12 | 1.03 (9.98) | 0.81 (10.55)
  Week 24: number analyzed (Participants) | 121 | 122
  Week 24 | 3.50 (11.05) | 1.39 (13.94)
  Week 36: number analyzed (Participants) | 110 | 110
  Week 36 | 3.21 (11.38) | 2.15 (13.42)
  Week 52: number analyzed (Participants) | 46 | 43
  Week 52 | 6.15 (13.87) | 3.09 (11.51)

8. Secondary Outcome: Time to First Acute Exacerbation of Idiopathic Pulmonary Fibrosis (IPF)
Time Frame: From Baseline up to 1 year
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Zinpentraxin Alfa | Placebo
Number analyzed (Participants) | 330 | 330
Months | NA [NA to NA] — NA = Not enough events available for estimation. | NA [NA to NA] — NA = Not enough events available for estimation.
Statistical Analysis 1: Comparison: Zinpentraxin Alfa; Test type: Superiority; p = 0.7005, Log Rank; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.40 to 1.86]

9. Secondary Outcome: Change in Carbon Monoxide Diffusing Capacity (DLCO)
Time Frame: At Baseline, Week 12, Week 24, Week 36 and Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: DLCO% Predicted
Arm/Group | Zinpentraxin Alfa | Placebo
Number analyzed (Participants) | 318 | 313
DLCO% Predicted
  Baseline | 51.73 (17.73) | 51.66 (14.78)
  Week 12: number analyzed (Participants) | 153 | 165
  Week 12 | -1.19 (11.89) | -2.78 (9.86)
  Week 24: number analyzed (Participants) | 110 | 108
  Week 24 | -4.68 (7.93) | -4.01 (9.75)
  Week 36: number analyzed (Participants) | 95 | 90
  Week 36 | -5.83 (8.49) | -4.66 (7.10)
  Week 52: number analyzed (Participants) | 32 | 36
  Week 52 | -6.30 (9.56) | -6.68 (9.28)

10. Secondary Outcome: Survival
Description: Survival is measured by all-cause mortality
Time Frame: From Baseline up to 1 year
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Zinpentraxin Alfa | Placebo
Number analyzed (Participants) | 330 | 330
Months | NA [NA to NA] — NA = Not enough events available for estimation. | NA [NA to NA] — NA = Not enough events available for estimation.

11. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Time Frame: From Baseline up to 8 weeks after the last dose of study drug (up to an average of 1 year)
Population: The safety population included all randomized participants who received at least one administration (full or partial dose) of study drug and were grouped according to the actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Zinpentraxin Alfa | Placebo
Number analyzed (Participants) | 331 | 329
Participants | 247 | 238

12. Secondary Outcome: Percentage of Participants With Infusion-related Reactions (IRRs) and Other Adverse Events of Special Interest
Time Frame: From Baseline up to 8 weeks after the last dose of study drug (up to an average of 1 year)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Zinpentraxin Alfa | Placebo
Number analyzed (Participants) | 331 | 329
Participants | 12 | 5

13. Secondary Outcome: Percentage of Participants Permanently Discontinuing Study Treatment Due to AEs
Time Frame: From Baseline up to 8 weeks after the last dose of study drug (up to an average of 1 year)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Zinpentraxin Alfa | Placebo
Number analyzed (Participants) | 331 | 329
Participants | 9 | 6

14. Secondary Outcome: Plasma Concentrations of PRM-151
Time Frame: Days 1, 5 and Weeks 4, 12, and 24
Population: The pharmacokinetic (PK) population included all randomized participants who received at least one administration (full or partial dose) of zinpentraxin alfa and at least one evaluable postdose PK sample that was above the lower limit of quantification (LLOQ).
Measure: Mean (Standard Deviation); unit: micrograms per millilitre (ug/mL)
Arm/Group | Zinpentraxin Alfa
Number analyzed (Participants) | 310
micrograms per millilitre (ug/mL)
  Day 1 -pre infusion: number analyzed (Participants) | 0
  Day 1 - 1h Post Infusion: number analyzed (Participants) | 33
  Day 1 - 1h Post Infusion | 198 (56.8)
  Day 1 - 2h Post Infusion | 203 (68.4)
  Day 1 - 4h Post Infusion: number analyzed (Participants) | 33
  Day 1 - 4h Post Infusion | 168 (48.0)
  Day 1 - 8h Post Infusion: number analyzed (Participants) | 15
  Day 1 - 8h Post Infusion | 118 (37.8)
  Day 1 - 10h Post Infusion: number analyzed (Participants) | 18
  Day 1 - 10h Post Infusion | 158 (35.8)
  Day 1 - 12h Post Infusion: number analyzed (Participants) | 15
  Day 1 - 12h Post Infusion | 95.9 (31.5)
  Day 1 - 24h Post Infusion: number analyzed (Participants) | 33
  Day 1 - 24h Post Infusion | 81.8 (26.2)
  Day 5 - Pre Infusion: number analyzed (Participants) | 303
  Day 5 - Pre Infusion | 39.6 (21.5)
  Day 5 - 2h Post Infusion: number analyzed (Participants) | 301
  Day 5 - 2h Post Infusion | 244 (75.6)
  Week 4 - Pre Infusion: number analyzed (Participants) | 276
  Week 4 - Pre Infusion | NA (NA) — NA = the drug level was below the limit of quantification of the assay.
  Week 4 - 2h Post Infusion: number analyzed (Participants) | 280
  Week 4 - 2h Post Infusion | 212 (105)
  Week 12 - Pre Infusion: number analyzed (Participants) | 180
  Week 12 - Pre Infusion | NA (NA) — NA = the drug level was below the limit of quantification of the assay.
  Week 12 - 2h Post Infusion: number analyzed (Participants) | 180
  Week 12 - 2h Post Infusion | 177 (72.7)
  Week 24 - Pre Infusion: number analyzed (Participants) | 133
  Week 24 - Pre Infusion | NA (NA) — NA = the drug level was below the limit of quantification of the assay.

15. Secondary Outcome: Prevalence of Anti-drug Antibodies (ADAs) at Baseline
Time Frame: At Baseline
Population: The immunogenicity population included all randomized participants with at least one postdose ADA assessment and were grouped according to treatment received or, if no treatment is received prior to study discontinuation, according to treatment assigned. There is no data reported for the Placebo Arm as that group never received any study drug. As such, we cannot measure anti-drug antibodies for that group of participants.
Measure: Number; unit: Participants
Arm/Group | Zinpentraxin Alfa
Number analyzed (Participants) | 255
Participants | 0

16. Secondary Outcome: Percentage of Participants With ADAs During the Study
Time Frame: Days 1, 5 and Weeks 4, 12, 24, 36, 48, 52 and 56
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Zinpentraxin Alfa
Number analyzed (Participants) | 280
Participants | 3

ADVERSE EVENTS:
Time Frame: From Baseline up to 8 weeks after the last dose of study drug (up to an average of 1 year)
Description: All-cause mortality was reported based on randomized population =all randomized participants.
  SAEs & other AEs reported based on safety-evaluable population which included all randomized participants who received at least one administration (full or partial dose) of study drug and were grouped according to the actual treatment received.
Arm/Group | Zinpentraxin Alfa | Placebo
All-Cause Mortality (participants affected / at risk) | 4/331 | 4/333
Serious Adverse Events (participants affected / at risk) | 46/331 | 40/329
Other Adverse Events (participants affected / at risk) | 140/331 | 128/329
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zinpentraxin Alfa (N=331) | Placebo (N=329)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (2) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric artery embolism (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 3 (3)
General physical health deterioration (General disorders) | 1 (1) | 1 (1)
Hernia (General disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2)
Device dislocation (Product Issues) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal embolism (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal infarct (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 8 (8)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Microscopic polyangiitis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zinpentraxin Alfa (N=331) | Placebo (N=329)
Diarrhoea (Gastrointestinal disorders) | 35 (48) | 34 (39)
Fatigue (General disorders) | 17 (22) | 14 (14)
COVID-19 (Infections and infestations) | 57 (59) | 57 (60)
Infusion related reaction (Injury, poisoning and procedural complications) | 31 (42) | 29 (55)
Cough (Respiratory, thoracic and mediastinal disorders) | 42 (46) | 38 (42)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 27 (29) | 20 (22)

LIMITATIONS AND CAVEATS:
This study was terminated early based on the futility analysis which concluded that zinpentraxin alfa was unlikely to meet its primary endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/99/NCT04552899/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/99/NCT04552899/SAP_001.pdf